CLINICAL TRIAL: NCT04295330
Title: Efficacy of Prolonging Intravenous Lidocaine by 72 Hours on Postoperative Pain and Recovery in Patients Undergoing Hepatectomy: a Prospective Randomized Controlled Study
Brief Title: Efficacy of Intravenous Lidocaine on Postoperative Pain and Recovery in Patients Undergoing Hepatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Chunling Jiang, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018HXFH046
Record Dates: First submitted 2020-02-16; First posted 2020-03-04 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Primary Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Lidocaine; Injections; Saline Solution

STUDY DESIGN:
Intervention Model Description: The experimental group received lidocaine and the control group received the same amount of saline.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participants, the anesthesiologist, data collectors, the physicians performing the follow-up, and data analysts will be blinded to the group allocation. Blinding will maintain until the completion of the final analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lidocaine group (Experimental): at the end of the induction of general anesthesia, a bolus injection of lidocaine 1.5 mg/kg, calculated using the patient's ideal body weight and given as an infusion over 10 minutes, followed by a continuous infusion of lidocaine at 1.5 mg/kg per hour for the whole surgical procedure and will be discontinued at the end of surgery.
  Interventions: Drug: Lidocaine Hydrochloride, Injectable
- placebo group (Placebo Comparator): the same volume of normal saline will be administered during anesthesia.
  Interventions: Drug: 0.9% normal saline

INTERVENTIONS:
Drug: Lidocaine Hydrochloride, Injectable — In the lidocaine group, at the end of the induction of general anesthesia, a bolus injection of lidocaine 1.5 mg/kg, calculated using the patient's ideal body weight and given as an infusion over 10 minutes, followed by a continuous infusion of lidocaine at 1.5 mg/kg per hour for the whole surgical procedure and will be discontinued at the end of surgery. Postoperative pain management during the first 72 postoperative hours will involve the use of a PCIA device, which will contain lidocaine 30mg/kg, sufentanil 2 μg/kg, granisetron 12 mg diluted to 200 mL in 0.9 % normal saline.
  Other Names: lidocaine group
  Arms: Lidocaine group
Drug: 0.9% normal saline — In the placebo group, the same volume of normal saline will be administered during anesthesia. The postoperative PCIA device will contain sufentanil 2 μg/kg, granisetron 12 mg diluted to 200 mL in 0.9% normal saline solution with a total volume of 200 ml.
  Other Names: placebo group
  Arms: placebo group

SUMMARY:
Patients who meet the enrollment criteria will be randomized 1:1 to either the lidocaine or the placebo group.

In the lidocaine group, at the end of the induction of general anesthesia, a bolus injection of lidocaine 1.5 mg/kg, calculated using the patient's ideal body weight and given as an infusion over 10 minutes, followed by a continuous infusion of lidocaine at 1.5 mg/kg per hour for the whole surgical procedure and will be discontinued at the end of surgery. In the placebo group, the same volume of normal saline will be administered during anesthesia.

DETAILED DESCRIPTION:
Patients who meet the enrollment criteria will be randomized 1:1 to either the lidocaine or the placebo group.

In the lidocaine group, at the end of the induction of general anesthesia, a bolus injection of lidocaine 1.5 mg/kg, calculated using the patient's ideal body weight and given as an infusion over 10 minutes, followed by a continuous infusion of lidocaine at 1.5 mg/kg per hour for the whole surgical procedure and will be discontinued at the end of surgery.

Blood samples will be drawn immediately after the bolus infusion of lidocaine, at the end of the surgery, and 24 hours after surgery to measure plasma lidocaine concentrations. Blood samples will also be collected 24 hours after surgery for subsequent measurement of IL-6, and tumor necrosis factor-α (TNF-α). The obtained samples will be labeled, centrifuged, frozen, and stored locally at -80° for subsequent testing.

Postoperative pain management during the first 72 postoperative hours will involve the use of a PCIA device, which will contain lidocaine 30mg/kg, sufentanil 2 μg/kg, granisetron 12 mg diluted to 200 mL in 0.9 % normal saline. In the placebo group, the same volume of normal saline will be administered during anesthesia. The postoperative PCIA device will contain sufentanil 2 μg/kg, granisetron 12 mg diluted to 200 mL in 0.9% normal saline solution with a total volume of 200 ml. All the background infusions of PCIA will set at 2 ml/h, the bolus volume of each PCIA press is 2 ml and the lockout interval is 15 min.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-80 years old
* American Society of Anesthesiologists(ASA) Ⅰ～III
* patients scheduled for elective hepatectomy

Exclusion Criteria:

• body weight < 40 kg or >100 kg; metastases occurring in other distant organs; severe hepatic insufficiency (aspartate aminotransferase or alanine transaminase or bilirubin > 2.5 times the upper limit of normal), renal impairment (creatinine clearance < 60 ml/min); cardiac rhythm disorders or systolic heart failure (second-and third-degree heart block, ejection fraction < 50%); with allergies to any of the trial drugs; inability to comprehend numeric rating scale.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-05-27 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the incidence of moderate to severe pain (NRS ≥ 4) during movement (i.e. deep breathing) at 24 hours after surgery. | The first 24 hours after surgery
  The pain is evaluated using numerical rating scale（NRS). NRS scores range from 0 to 10 points, with 0 points representing no pain, 1-3 points representing mild pain, 4-6 points representing moderate pain, 7-9 points representing severe pain and 10 points representing the strongest pain.

SECONDARY OUTCOMES:
The incidence of moderate to severe pain at 24 hours after surgery at rest | The first 24 hours after surgery
  The pain is evaluated using numerical rating scale（NRS). NRS scores range from 0 to 10 points, with 0 points representing no pain, 1-3 points representing mild pain, 4-6 points representing moderate pain, 7-9 points representing severe pain and 10 points representing the strongest pain.
The incidence of moderate to severe pain at 48 and 72 hours after surgery at rest and during movement; | At 3 days after surgery
  The pain is evaluated using numerical rating scale（NRS). NRS scores range from 0 to 10 points, with 0 points representing no pain, 1-3 points representing mild pain, 4-6 points representing moderate pain, 7-9 points representing severe pain and 10 points representing the strongest pain.
The cumulative morphine consumption at 24, 48 and 72 hours postoperatively | At the end of the surgery，24，48 and 72 hours after surgery
  intra-operative and postoperative opioid use is reported as morphine milligram equivalents, calculated using the Practical Pain Management calculator
Bowel function recovery | At 3 days after surgery
  defined as the time to first defecation or time to first flatus
The incidence of PONV during the first 72 hours after surgery | At 3 days after surgery
  we considered it PONV if patients felt any nausea or had any vomiting
The incidence of a composite of postoperative pulmonary complications during hospitalization | during the period from the end of surgery to discharge
  defined as positive if any component developed before discharge after surgery; These complications included respiratory infection, respiratory failure, pleural effusion, atelectasis, pneumothorax, bronchospasm, or aspiration pneumonitis loading dose, immediately after the end of surgery, and at the first 24 hours after surgery
Length of hospital stay | during the period from the end of surgery to discharge
  determined by the number of days from admittance to discharge
Patient satisfaction scores | 72 hours after surgery and before discharge
  (satisfaction scores regarding pain control and the overall recovery process were obtained at 72 hours after surgery, using a 11-point Likert scale, with 0 indicating "very dissatisfied"and10 indicating "very satisfied"
Levels of inflammatory factors ( IL-6, TNF-α) at 24 hours after surgery. | at 24 hours after surgery.
  Levels of inflammatory factors ( IL-6, TNF-α) at 24 hours after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Chunling Jiang, PhD, Study Director — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu Y, Ye M, Liu F, Hong Y, Kang Y, Li Y, Li H, Xiao X, Yu F, Zhou M, Zhou L, Jiang C. Efficacy of prolonged intravenous lidocaine infusion for postoperative movement-evoked pain following hepatectomy: a double-blinded, randomised, placebo-controlled trial. Br J Anaesth. 2023 Jul;131(1):113-121. doi: 10.1016/j.bja.2023.03.026. Epub 2023 May 16. PMID 37202261